CLINICAL TRIAL: NCT02681601
Title: Nutrition Support to Improve Outcomes in Patients With Unresectable Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Do Well Laboratories Inc. (Unknown); Hirshberg Foundation for Pancreatic Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-001926
Record Dates: First submitted 2016-01-27; First posted 2016-02-12 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2021-10

CONDITIONS: Cancer of Pancreas
Keywords: Diet, Food, and Nutrition
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet + Nutrawell Powder with Fish Oil (Active Comparator): Subjects will be evaluated by a registered dietitian with a diet prescription (55% carbohydrate, 30% fat and 15% protein) including Nutrawell powder with fish oil.
  Interventions: Dietary Supplement: Nutrawell Powder; Dietary Supplement: OmegaRich fish oil supplement
- Dietary Intervention Only (Active Comparator): Subjects will be evaluated by a registered dietitian with a diet prescription (55% carbohydrate, 30% fat and 15% protein) not including servings of Nutrawell powder with fish oil.
  Interventions: Other: Diet Only

INTERVENTIONS:
Dietary Supplement: Nutrawell Powder — The NutraWell nutrition powder will be provided by and distributed from New Health Nutraceuticals (Irvine, California - USA). Nutrawell is manufactured New Health Enterprises, Inc. The supplement sample will be stored at room temperature in the UCLA Center for Human Nutrition research unit.
  OmegaRich Contains high concentration and high purity of natural omega-3 polyunsaturated fatty acids: Eicosapenatenoic acid (EPA) and docosahexaenoic acid (DHA) from deep water fish.
  Enriched with natural vitamin E: d- tocopherol Triglyceride form (TG-form) of the raw fish oil ingredients. Each fish oil capsule contains 55% EPA and DHA with 330 mg EPA and 220 mg DHA.
  Arms: Diet + Nutrawell Powder with Fish Oil
Other: Diet Only — Subjects will be evaluated by a registered dietitian and randomized to diet prescription (55% carbohydrate, 30% fat and 15% protein)
  Arms: Dietary Intervention Only
Dietary Supplement: OmegaRich fish oil supplement — OmegaRich is manufactured New Health Enterprises, Inc. The supplement sample will be stored at room temperature in the UCLA Center for Human Nutrition research unit.
  OmegaRich Contains: high concentration and high purity of natural omega-3 polyunsaturated fatty acids: Eicosapenatenoic acid (EPA) and docosahexaenoic acid (DHA) from deep water fish.
  Enriched with natural vitamin E: d- tocopherol Triglyceride form (TG-form) of the raw fish oil ingredients. Each fish oil capsule contains 55% EPA and DHA with 330 mg EPA and 220 mg DHA.
  Arms: Diet + Nutrawell Powder with Fish Oil

SUMMARY:
There are few well-designed studies evaluating the effect of nutrition support in patients with cancer cachexia. The aim of this study is to examine the effect of dietary prescription with and without nutrition supplementation in patients with unresectable pancreatic cancer on body weight, body composition, total calorie intake, quality of life and blood inflammatory markers.

DETAILED DESCRIPTION:
A total of 60 subjects will be recruited from The University of California Los Angeles (UCLA) Hirshberg Pancreatic Cancer Center, print and/or radio advertisements, UCLA campus wide e-mail, and flyers posted on campus and in the community. Participants will be pre-screened over the telephone to determine eligibility. Eligible subjects will be asked to come to the Center for Human Nutrition for a Screening Visit.

At screening, informed consent and authorization will be reviewed and signed a medical history will be obtained. The subjects will be screened by medical history/physical exam, a fasting blood sample will be collected for a comprehensive metabolic panel, a complete blood count, chemistry and liver function tests.

Day 1 will be the first study day. Subjects will come to the UCLA Center for Human Nutrition in the fasting state and remain for approximately ~1 hour. The food intake record will be collected and entered into the Automated Self- Administered Food Recall (NIH ASA24). The vital signs, anthropometric assessments will be measured and quality of life questionnaire will be completed.

A fasting blood sample (20 ml) will be collected for metabolic panel and inflammatory markers. A 6-minute walk will be done at the research center.

Subjects will be evaluated by a registered dietitian and randomized to diet prescription (55% carbohydrate, 30% fat and 15% protein) vs. the same diet prescription including three servings of supplement powder and fish oil. The research dietitian will develop meal plans based on basal metabolic rate and physical activity. Subjects will be provided a pedometer to wear daily. Any subject in either group who develops symptoms of pancreatic insufficiency will be provided with pancreatic enzyme supplementation.

Day 28, 56, 84 and 112 will be follow-up visits. The same procedures will be performed as on day 1. Subjects will come to the UCLA Center for Human Nutrition in the fasting state and remain for approximately ~1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable pancreatic adenocarcinoma
* Weight loss of greater than 5% in the previous 6 months
* Life expectancy of greater than 3 months and a Karnofsky performance score of 60 or more.
* Non-smokers

Exclusion Criteria:

* Chemotherapy other than gemcitabine
* Radiotherapy, or surgical treatment in the previous month
* Consumption of dietary supplements or medications such as steroids that could affect metabolism.
* Presence of ascites
* Liver function test > 2 standard deviation of upper limit
* Chronic or acute renal insufficiency
* Severe anemia with hemoglobin<10
* Uncontrolled pain
* Uncontrolled nausea and vomiting
* Participation in a therapeutic research study within 30 days of baseline
* Diet restrictions including vegetarianism and veganism
* Allergy or intolerance to fish and/or fish oil

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurement: Weight | At each visit outlined for 3 months
  Weight in Kilograms
Anthropometric measurement: Body Composition | At each visit outlined for 3 months
  Body Composition: kilogram weight of lean body mass

SECONDARY OUTCOMES:
Blood biochemistry | At each visit outlined for 3 months
  complete blood count
Blood biochemistry | At each visit outlined for 3 months
  Blood electrolytes
Blood biochemistry | At each visit outlined for 3 months
  Liver function test
Blood biochemistry | At each visit outlined for 3 months
  Lipid panel
Blood biochemistry | At each visit outlined for 3 months
  Pancreatic tumor markers
Blood biochemistry | At each visit outlined for 3 months
  Inflammatory markers
Physical activity | At each visit outlined for 3 months
  All subjects will be provided a pedometer to record daily steps.
Physical activity | At each visit outlined for 3 months
  A 6 minute walk will be done at each visit.
Physical activity | At each visit outlined for 3 months
  Karnofsky performance score
Quality of life: General | At each visit outlined for 3 months
  Measured with short form health survey (SF36)
Quality of life: Appetite | At each visit outlined for 3 months
  Appetite will be measured on a numerical rating scale between 0 and 10, where 0 indicated absolutely no appetite and 10 indicated an extremely good appetite (Simons et al, 1996)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Medicine Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lillemoe KD. Palliative therapy for pancreatic cancer. Surg Oncol Clin N Am. 1998 Jan;7(1):199-216. PMID 9443996
- [Background] Capra S, Bauer J, Davidson W, Ash S. Nutritional therapy for cancer-induced weight loss. Nutr Clin Pract. 2002 Aug;17(4):210-3. doi: 10.1177/0115426502017004210. PMID 16214989
- [Background] Stratton RJ. Should food or supplements be used in the community for the treatment of disease-related malnutrition? Proc Nutr Soc. 2005 Aug;64(3):325-33. doi: 10.1079/pns2005439. PMID 16048664
- [Background] Fearon KC, Von Meyenfeldt MF, Moses AG, Van Geenen R, Roy A, Gouma DJ, Giacosa A, Van Gossum A, Bauer J, Barber MD, Aaronson NK, Voss AC, Tisdale MJ. Effect of a protein and energy dense N-3 fatty acid enriched oral supplement on loss of weight and lean tissue in cancer cachexia: a randomised double blind trial. Gut. 2003 Oct;52(10):1479-86. doi: 10.1136/gut.52.10.1479. PMID 12970142
- [Background] Cawood AL, Elia M, Stratton RJ. Systematic review and meta-analysis of the effects of high protein oral nutritional supplements. Ageing Res Rev. 2012 Apr;11(2):278-96. doi: 10.1016/j.arr.2011.12.008. Epub 2011 Dec 22. PMID 22212388
- [Background] Goldberg MF, Custis PH. Retinal and other manifestations of incontinentia pigmenti (Bloch-Sulzberger syndrome). Ophthalmology. 1993 Nov;100(11):1645-54. doi: 10.1016/s0161-6420(93)31422-3. PMID 8233390
- [Background] Kraft M, Kraft K, Gartner S, Mayerle J, Simon P, Weber E, Schutte K, Stieler J, Koula-Jenik H, Holzhauer P, Grober U, Engel G, Muller C, Feng YS, Aghdassi A, Nitsche C, Malfertheiner P, Patrzyk M, Kohlmann T, Lerch MM. L-Carnitine-supplementation in advanced pancreatic cancer (CARPAN)--a randomized multicentre trial. Nutr J. 2012 Jul 23;11:52. doi: 10.1186/1475-2891-11-52. PMID 22824168
- [Background] Donohoe CL, Ryan AM, Reynolds JV. Cancer cachexia: mechanisms and clinical implications. Gastroenterol Res Pract. 2011;2011:601434. doi: 10.1155/2011/601434. Epub 2011 Jun 13. PMID 21760776
- [Background] Kleponis J, Skelton R, Zheng L. Fueling the engine and releasing the break: combinational therapy of cancer vaccines and immune checkpoint inhibitors. Cancer Biol Med. 2015 Sep;12(3):201-8. doi: 10.7497/j.issn.2095-3941.2015.0046. PMID 26487965
- [Background] Simons JP, Aaronson NK, Vansteenkiste JF, ten Velde GP, Muller MJ, Drenth BM, Erdkamp FL, Cobben EG, Schoon EJ, Smeets JB, Schouten HC, Demedts M, Hillen HF, Blijham GH, Wouters EF. Effects of medroxyprogesterone acetate on appetite, weight, and quality of life in advanced-stage non-hormone-sensitive cancer: a placebo-controlled multicenter study. J Clin Oncol. 1996 Apr;14(4):1077-84. doi: 10.1200/JCO.1996.14.4.1077. PMID 8648360